CLINICAL TRIAL: NCT02394951
Title: Investigation of Somatosensory Predictors of Response to Pregabalin in Painful Chemotherapy-induced Peripheral Neuropathy (CIPN)
Brief Title: Pregabalin in CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor, Department of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 201501067
Record Dates: First submitted 2015-03-04; First posted 2015-03-20 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Neuropathy; Pain
Keywords: chemotherapy
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Experimental): Pregabalin administered for 4 weeks, titrated to highest tolerated dose up to 600 mg/day.
  Interventions: Drug: Pregabalin; Drug: Placebo
- Placebo (Placebo Comparator): Identical, matching inactive substance administered for 4 weeks following the same dosing regimen.
  Interventions: Drug: Pregabalin; Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Anticonvulsant
  Other Names: Lyrica
Drug: Placebo — Identical, matching inactive substance

SUMMARY:
The investigators seek to investigate certain patient characteristics that would predict the response to a currently approved analgesic, pregabalin, in patients with chronic pain due to nerve damage caused by chemotherapy. Patients with this painful condition, called chemotherapy-induced peripheral neuropathy (CIPN) have a current or recent history of chemotherapy with particular chemotherapy agents called taxanes or oxaliplatin. The investigators will recruit potential subjects from both the Siteman Cancer Center and the Washington University Pain Management Center. Those patients who meet the inclusion and satisfy the exclusion criteria will be enrolled. Subjects will undergo mechanical and thermal sensitivity testing on their extremities, will provide quality of life information by completing questionnaires and will receive pregabalin followed by placebo, or placebo followed by pregabalin [crossover design] in order to assess how well the sensory tests predict the analgesic effect of pregabalin (compared to placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Distal symmetric pain distribution (both feet, with or without pain in hands).
3. The pain appeared during or up to 12 weeks after treatment with oxaliplatin, paclitaxel, docetaxel or any combination of these.
4. Score of 4 or more on DN4 (Douleur Neuropathique 4) neuropathic pain questionnaire
5. Pain duration > 2 months.
6. Patient report of average daily pain intensity in the last week >3 on 0-10 Numerical Rating Scale (NRS).
7. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation.
8. Able and willing to sign an IRB-approved written informed consent.

Exclusion Criteria:

1. Hypersensitivity to pregabalin.
2. Current treatment with pregabalin.
3. Current treatment with a vinca alkaloid (e.g. vincristine, vinblastine), or CIPN that may be associated with previous treatment with a vinca alkaloid.
4. History of diabetes mellitus or a neurological disorder with any previous signs of distal symmetric polyneuropathy.
5. Moderate to severe renal failure (Creatinine clearance < 30mL/min, by Cockcroft-Gault formula).
6. ALT (alanine aminotransferase) or AST (aspartate aminotransferase ) > 3 times the upper limit of normal.
7. Planned surgeries or radiation treatment within 10 weeks following study inclusion.
8. Inability to complete pain self-report.
9. Pregnancy or lactation
10. Patients with seizure disorders treated with anticonvulsants
11. Current participation in a trial with another investigational agent.
12. Concomitant medication as follows:

    * Subjects treated with gabapentin or other anticonvulsant for neuropathic pain will be required to taper the medication and discontinue for at least 2 weeks prior to study initiation.
    * Patients on antidepressant treatment for pain or depression (TCAs, SSRI, SNRIs etc. will be allowed to continue their medications provided they have been on a stable dose for at least 4 weeks before study initiation. No dose regimen changes of antidepressants will be allowed during the study period.
    * Patients on around-the clock opioid treatment (including tramadol) will be allowed to continue their medication provided they have been on a stable dose for at least 4 weeks before study initiation. The maximum allowed dose of opioid will be equivalent to 60mg oral morphine sulphate. Patients with higher doses will be required to taper down their opioid dose to maximum 60mg oral morphine equivalent, and continue on stable dose for 4 weeks before enrollment in the study. Short-acting opioids for painful CIPN treatment will not be allowed.
    * Treatment with non-steroidal anti-inflammatory drugs (NSAIDs) will be discontinued at least 2 weeks before study initiation. However, low-dose aspirin (≤325mg/day) will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin First Then Placebo: Pregabalin administered for 4 weeks, titrated to highest tolerated dose up to 600 mg/day.
  Pregabalin: Anticonvulsant
  Placebo: Identical, matching inactive substance
- Placebo First Then Pregabalin: Identical, matching inactive substance administered for 4 weeks following the same dosing regimen.
  Pregabalin: Anticonvulsant
  Placebo: Identical, matching inactive substance
Period: Period I
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 12 | 14
Completed | 11 | 13
Not Completed | 1 | 1
Period: Period II
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 11 | 13
Completed | 11 | 9
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.2) | 59.9 (11.4) | 62.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 10 | 14 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Spontaneous Pain Intensity as a Function of Baseline MPT
Description: Correlation between Mechanical Pain Threshold (MPT in mN) at baseline and reduction in spontaneous pain intensity (% reduction on 0-10 NRS) at the end of 4-week treatment. The slopes (Pearson coefficients) of the correlation obtained from pregabalin vs. placebo will be compared.
Time Frame: Baseline to week 4
Measure: Number (95% Confidence Interval); unit: Pearson correlation coefficient
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 23
Pearson correlation coefficient | -0.0179 [-0.0459 to 0.0101] | -0.0172 [-0.0514 to 0.0170]

2. Secondary Outcome: Absolute Change in Pain Intensity, Measured on 0-10 Numerical Rating Scale (NRS)
Description: Absolute change in pain intensity on 0-10 numerical rating scale (NRS) from baseline to 4 weeks with pregabalin vs. placebo NRS: 0= no pain, 10= worst pain
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 NRS)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale (0-10 NRS) | -1.0 (1.13) | 0.3 (1.10)

3. Secondary Outcome: Change in NPSI Outcomes
Description: Change from baseline to week 4 in total NPSI (Neuropathic Pain Symptom Inventory) score The total NPSI score is comprised by adding 5 sub-scores (Burning pain, Pressing pain, Paroxysmal pain, Evoked pain, and Paresthesia/Dysesthesia) and is expressed on a 0-100 scale; 0-minimum (least), and 100 maximum (worst) score
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: units on a scale (0-100 NPSI score)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale (0-100 NPSI score) | -9.8 (12.49) | 1.8 (20.93)

4. Secondary Outcome: Change in BPI Outcomes (SEVERITY)
Description: Change from baseline to week 4 in BPI (Brief Pain Inventory) pain severity severity score BPI severity score is expressed on 0-10 scale, with 0 being the minimum (least), and 10 being the maximum (worst) pain severity
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 BPI severity)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale (0-10 BPI severity) | -0.8 (1.52) | -0.1 (1.14)

5. Secondary Outcome: Change in Sleep Problem Index (SPI) Outcomes
Description: Change from baseline to week 4 in SPI (Sleep Problem Index) score, on 0-100 scale, where 0= best (least) score, and 100= maximum (worst) score
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: units on a scale (0-100 SPI)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale (0-100 SPI) | -5.1 (9.45) | -4.1 (11.64)

6. Secondary Outcome: Change in BPI Outcomes (INTERFERENCE)
Description: Change from baseline to week 4 in BPI (Brief Pain Inventory) pain interference score BPI interference score is expressed on 0-10 scale, with 0 being the minimum (least), and 10 being the maximum (worst) pain interference
Time Frame: baseline to week 4
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 BPI interference)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale (0-10 BPI interference) | -0.6 (1.64) | -0.2 (1.10)

7. Secondary Outcome: Number of Patients With Significant Pain Reduction
Description: Number of patients who experienced 50% or more reduction in average daily pain (on 0-10 NRS, Numerical Rating Scale, where 0=least pain, 10=worst pain)
Time Frame: Baseline to week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 11 weeks
Description: Common Terminology Criteria for Adverse Events - CTCAE version 4.0
Arm/Group | Pregabalin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=25) | Placebo (N=25)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Small bowel obstruction in the setting of a new oncological diagnosis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=25) | Placebo (N=25)
Dizziness (Nervous system disorders) | 17 | 4
Somnolence (Nervous system disorders) | 22 | 11
Dry Mouth (Gastrointestinal disorders) | 14 | 10
Edema (General disorders) | 8 | 8
Weight Gain (Investigations) | 4 | 1
Headache (Nervous system disorders) | 10 | 11
Nausea (Gastrointestinal disorders) | 6 | 7
Blurred Vision (Eye disorders) | 8 | 4
Gait Disturbance (General disorders) | 2 | 0
Spasticity (Nervous system disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Early termination due to slow recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT02394951/Prot_SAP_000.pdf